CLINICAL TRIAL: NCT00524940
Title: Immunogenicity and Safety of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2007-2008 Formulation (Intramuscular Route)
Brief Title: Trial to Describe the Safety and Immunogenicity of Fluzone®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRC37
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Results first posted 2009-03-30 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza; Orthomyxoviruses; Inactivated Split-virion influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: Inactivated, Split-Virion Influenza Virus

INTERVENTIONS:
Biological: Inactivated, Split-Virion Influenza Virus — 0.5 mL, Intramuscular
  Other Names: Fluzone®

SUMMARY:
Objective 1:To describe the safety of the inactivated, split-virion influenza vaccine, Northern Hemisphere (NH) 2007-2008 formulation.

Objective 2: To describe the immunogenicity, of Fluzone, inactivated, split virion influenza vaccine NH 2007-2008 formulation.

Objective 3: Serum Collection - To submit remaining available sera to Center for Biologics Evaluation and research (CBER) for further analysis by the Food and Drug Administration (FDA), the Center for Disease Control and Prevention (CDC), and the World Health Organization (WHO) to support selection and recommendation of antigen strains for subsequent influenza vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years or older on the day of inclusion.
* Participant able to attend scheduled visits and to comply with the study procedures during the entire duration of the study.
* Participant is in good health as assessed by the investigator.
* Participant willing and able to meet protocol requirements.
* Participant willing and able to give informed consent.
* For a woman, inability to bear a child or negative serum/urine pregnancy test.

Exclusion Criteria:

* Self-reported allergy to egg proteins, chicken proteins, or one of the constituents of the vaccine, such as thimerosal or formaldehyde.
* An acute illness with or without fever (temperature ≥ 99.5 °F oral) in the 72 hours preceding enrollment in the trial.
* Clinically significant findings in vital signs (including temperature ≥ 99.5 °F oral) on review of systems.
* Self-reported history of severe adverse event to any influenza vaccine.
* Laboratory-confirmed influenza infection or vaccination against influenza in the 6 months preceding enrollment in the study.
* Any vaccination in the 14 days preceding enrollment in the study or scheduled between Visit 1 and Visit 2.
* Participation in any other interventional drug or vaccine trial within the 30 days preceding or during enrollment into this study.
* Immunocompromising or immunosuppressive therapy (including systemic steroid use for 2 weeks or more), cancer chemotherapy, or radiation therapy at the time of enrollment, planned during the period of this study, or at any time within the past 6 months.
* Receipt of blood or blood products within the 3 months preceding enrollment in the study.
* Diabetes mellitus requiring pharmacological control.
* Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Person deprived of freedom by an administrative or court order (having legal or medical guardian).
* For women of childbearing potential, a positive urine pregnancy test, breast feeding, or not using a medically approved form of contraception for the duration of the trial.
* Current alcohol or drug use that may interfere with the subject's ability to comply with trial procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Prior personal history of Guillain-Barré syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc
Locations (1):
- Norfolk, Virginia, United States

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 15 August to 24 September 2007 at one US clinic site.
Pre-assignment Details: A total of 124 participants that met the inclusion and exclusion criteria were enrolled and vaccinated.
Groups:
- Study Group: All participants enrolled and received Fluzone® Vaccine
Period: Overall Study
Arm/Group | Study Group
Started | 124
Completed | 124
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 124
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.40 (19.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 124

OUTCOME MEASURES:

1. Primary Outcome: Solicited Injection Site and Solicited Systemic Reactions Post-vaccination.
Description: Information concerning the safety of Fluzone® vaccine 2007-2008 formulation.
Time Frame: 0-3 days post-vaccination and entire study duration
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat Population.
Measure: Number; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 124
Participants
  Any Solicited Injection Site Reaction | 62
  Any Pain | 57
  Grade 3 Pain (Incapacitating) | 0
  Any Redness | 9
  Grade 3 Redness (≥5.0 cm) | 0
  Any Swelling | 7
  Grade 3 Swelling (≥ 5.0 cm) | 1
  Any Induration | 8
  Grade 3 Induration (≥ 5.0 cm) | 0
  Any Ecchymosis | 5
  Grade 3 Ecchymosis (≥ 5.0 cm) | 0
  Any Solicited Systemic Reaction | 40
  Any Fever | 3
  Grade 3 Fever (> 102.2°F) | 0
  Any Headache | 26
  Grade 3 Headache (Prevented daily activities) | 1
  Any Malaise | 15
  Grade 3 Malaise (Prevented daily activities) | 0
  Any Myalgia | 27
  Grade 3 Myalgia (Prevented daily activities) | 0
  Any Shivering | 1
  Grade 3 Shivering (Prevented daily activities) | 0

2. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition Antibodies Pre-vaccination and Post-vaccination.
Description: GMTs and their 95% Confidence Interval are presented for each of the 3 antigens in the Fluzone® Vaccine 2007-2008 formulation.
Time Frame: 21 days post-vaccination
Population: The GMT were evaluated in the per-protocol Population
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Study Group
Number analyzed (Participants) | 112
Titer
  H1N1 A/Solomon Islands/3/2006 - PRE | 30.7 [23.4 to 40.2]
  H1N1 A/Solomon Islands/3/2006 - POST | 234.1 [180.6 to 303.5]
  H3N2 A/Wisconsin/67/2005 - PRE | 88.1 [66.7 to 116.2]
  H3N2 A/Wisconsin/67/2005 - POST | 347.9 [281.0 to 430.7]
  B/Malaysia/2506/2004 - PRE | 13.0 [11.0 to 15.4]
  B/Malaysia/2506/2004 - POST | 35.9 [29.4 to 43.8]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to 21 days post-vaccination.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/124
Other Adverse Events (participants affected / at risk) | 57/124
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group (N=124)
Injection site pain (General disorders) | 57
Injection site redness (General disorders) | 9
Injection site swelling (General disorders) | 7
Injection site induration (General disorders) | 8
Headache (Nervous system disorders) | 26
Malaise (General disorders) | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.